CLINICAL TRIAL: NCT06640985
Title: A Single-center Prospective Case Series Study to Determine the Efficacy and Safety of EDX110 in Hard-to-heal Wounds Resulting From Venous Insufficiency or Diabetes
Brief Title: EDX110 - Efficacy and Safety in the Management of Hard-to-heal Wounds
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WC-24-446
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Wound Healing; Diabetic Foot; Foot Ulcer, Diabetic; Venous Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic Foot Ulcer (DFU) (Experimental): DFU treatment with EDX110 wound dressing
  Interventions: Device: EDX110 wound dressing system
- Venous Leg Ulcer (VLU) (Active Comparator): VLU treatment with EDX110 wound dressing
  Interventions: Device: EDX110 wound dressing system

INTERVENTIONS:
Device: EDX110 wound dressing system — EDX110 is a dressing system comprising two layers that allows the generation of nitric oxide (NO) in situ, enables adequate moisture management and facilitates debridement

SUMMARY:
Post-market study to determine the efficacy of EDX110 dressing system in hard-to-heal wounds.

DETAILED DESCRIPTION:
Prospective, single-center, non-blinded, non-randomized, post-market study to determine the efficacy of EDX110 dressing system in diabetic foot ulcers (DFUs) and venous leg ulcers (VLUs).

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years old and willing to participate in all procedures and follow-up evaluations necessary to complete the study
* An index ulcer meeting the following characteristics:

  * Diabetic foot ulcer (DFU): Wagner Grade 1: partial- or full-thickness (superficial)
  * DFU: Located on the anatomical foot; defined as distal to the medial malleolus
  * Venous leg ulcer (VLU): Partial or full thickness
  * VLU: Located below the knee and above the ankle
  * Presents with or without clinical signs of superficial infection
  * Present for ≥4 weeks and <52 weeks
  * Wounds will be dry to moderately exudating
  * Post-debridement wound area is ≥0.5 cm2 and ≤25 cm2
* If two or more ulcers are present, the index ulcer must additionally be:

  * The ulcer with the largest wound area
  * ≥3cm distance from any other ulcer on the affected limb
* DFU: type 1 or type 2 diabetes (confirmed by the subject's medical history)
* DFU: HgbA1c <9% at screening
* GFR>30 mL/min/1,73m2
* Subject has adequate circulation to the affected extremity, as demonstrated by at least one of the following results within the past 30:

  * Dorsum transcutaneous oxygen test (TcPO2): >30mmHg;
  * Subject's Ankle-Brachial Index (ABI) by Doppler: ≥0.7 and ≤1.2;
  * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of the affected foot. For Ankle-Brachial Pressure Index (ABPI): >1.2, for Toe Brachial Index (TBI): >0.5
* A total lymphocyte count of more than 1500 cells/mm3
* Albumin level of more than 3.5 g/dL
* Subject can ambulate at home or in the clinic with or without mobility aids
* BMI ≤45

Exclusion Criteria:

* Subjects with wounds that have any of the following characteristics:

  • Wounds that penetrate down to tendon, ligament, joint capsule or bone, underlying muscle tissue, or organs
* Tunnelling wounds

  * Known or suspected local skin malignancy at the site of the ulcer
  * DFU: Major structural abnormalities of the foot
  * DFU: Active Charcot deformity
  * VLU: inability to tolerate elastocompression (40 mm/hg)
  * Wound duration >1 year
* Subjects receiving any of the following prior therapies:

  * In the last 10 days:

    * Chemical debridement
    * Dakin's solution
    * Medical honey therapy
  * In the last 30 days (or anticipated to require such medications during the study period):

    * Cytotoxic chemotherapy
    * Application of topical steroids to the ulcer surface
    * Use of ≥14 days of immune suppressants (including systemic corticosteroids) OR
    * Subject is anticipated to require such medications during the study period
  * In the last 30 days:

    o Study ulcer treatment with any advanced therapy, including, biomedical or topical growth factors, tissue engineered materials
  * In the last 6 months:

    * Any amputation to the affected leg
    * Revascularization (surgical or stenting) to the affected leg
* Known hypersensitivity to constituents of the product
* Osteomyelitis/bone infection of the affected foot/leg, as verified by x-ray within 30 days prior to screening
* Active cellulitis at the wound site
* History of radiation at the ulcer site, regardless of duration
* Chronic kidney disease stage 4 or 5
* Immune system disorders, including SLE, AIDS or HIV
* Presence of any other pathology that would limit blood supply and compromise healing
* Revascularization procedure to increase blood flow in the target limb
* Presence of any condition (including current drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of, or compliance with the study
* Women of childbearing age (women aged <55 years who have not undergone menopause) who are:

  * Pregnant at time of enrolment
  * Planning to become pregnant during the time of the study
  * Have been pregnant within the last 6 months
  * Breast-feeding
  * Unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence) during the time of the study
  * Concurrent enrolment in any other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Effect of EDX110 in reducing the wound size of commonly occurring hard-to-heal wounds: DFUs and VLUs | 12 week
  Percentage area reduction (PAR) of target wound at 12 weeks for each wound determined by wound measurements

SECONDARY OUTCOMES:
Efficacy of EDX110 in complete wound management and healing of hard-to-heal wounds | 4 week
  PAR of target wound as defined as 100% reepithelialization
Effect of EDX110 | Treatment, week 4 and 12
  Treatment effect by using the 17-item Wound Quality of Life (W-QoL) questionnaire, assessing how wound care has affected the quality of life in the last seven days, ranging from "Not at all" to "Very much"
Tolerability of EDX110 | up to 12 week
  Tolerability assessed by Visual Analog Scale (VAS), assessing overall impression and satisfaction, ranging from "Very Poor" to "Excellent"

OTHER OUTCOMES:
Complications | up to 12 week
  Number and type of wound and device-related Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Jeison David Peñuela, MD, Principal Investigator — Convatec Medical Care
Locations (1):
- Convatec Medical Care, Santiago, Chile